CLINICAL TRIAL: NCT04252599
Title: Upper Airway Function and Cardiorespiratory Performance in Impair Trunk Motor Control Multiple Sclerosis Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, assistant professor, Universidad de Granada
Other Study IDs: DF0088UG
Record Dates: First submitted 2020-01-23; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group
- Multiple sclerosis group
- Multiple sclerosis trunk impairment

SUMMARY:
Multiple sclerosis is a chronic and highly disabling disorder with considerable social impact and economic consequences. It is caused by damage to the myelin sheath, the protective covering that surrounds nerve cells. Different areas are affected, including upper airway function, trunk motor control and cardiorespiratory performance. The aim of this study was to determinate the relevance of trunk motor control in upper airway function and cardiorespiratory performance in patients with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of MS in any of its forms according to McDonald criteria
* Were aged higher than 18 years
* No pathology in the uppers extremities
* Capacity to understand and response the questionnaires
* Ability to provide informed consent.

Exclusion Criteria:

* Cancer diagnoses, cognitive or psychiatric disorders, severe musculoskeletal disorders, severe orthopaedic problems, organ failure, incapacity to cooperate
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Have a diagnosis of MS in any of its forms according to McDonald criteria
  * Were aged higher than 18 years
  * No pathology in the uppers extremities
  * Capacity to understand and response the questionnaires
  * Ability to provide informed consent.
  Exclusion Criteria:
  * Cancer diagnoses, cognitive or psychiatric disorders, severe musculoskeletal disorders, severe orthopaedic problems, organ failure, incapacity to cooperate
  * Inability to provide informed consent.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2020-01-24 (Estimated)

PRIMARY OUTCOMES:
Trunk motor control | baseline
  The impairment of trunk motor control was measured with the Modified Trunk Impairment Scale (mTIS). The values range to 0 from 16 being higher values, better trunk motor control.
Swallowing function | baseline
  To evaluate swallowing function we used two questionnaires: the Swallowing quality of life questionnaire (SWAL-QOL). It contains 44 items and each item was scored from zero (the worst state) to four (the best state).
Swallowing function | baseline
  To evaluate swallowing function we used two questionnaires: the Eating Assessment Tool-10 (EAT-10). The values range from 0 to 4 being higher values worse swallowing function.
Ventilation function | baseline
  Ventilation capacity was measured with spirometry and peak flow using Spirobank II (MIR, Italy).
Phonation function | baseline
  The phonatory function and it´s repercussion on daily life was evaluated by the Voice handicap index (VHI-30),
The exercise capacity focussed on lower limbs | baseline
  The Five-Times-Sit-to-Stand test (5STS)
The exercise capacity focussed on upper limbs | baseline
  The exercise capacity focussed on upper limbs was measured by the unsupported upper-limb exercise test (UULEX)
The anaerobic threshold | baseline
  Incremental sit-to-stand test (ISTS)

SECONDARY OUTCOMES:
Psychological status | baseline
  Psychological status was evaluated with and the Beck Depression Inventory (Beck) to measure depression. The values range to 0 from 63, being higher values, most severe depression.
Psychological status | baseline
  Psychological status was evaluated with the Beck Anxiety Inventory (BAI) to measure anxiety. The values range to 0 from 63, being higher values, most severe anxiety.
The degree of neurological functioning | baseline
  The degree of neurological functioning in patients with MS was measured with the Kurtzke Expanded Disability Status Scale (EDSS). The values range to 0 from 10, being 0 normal status healthy and 10 the death.
The impact of the multiple sclerosis disease | baseline
  The impact of the disease was determinate with the Multiple Sclerosis Impact Scale (MSIS-29).
  It´s an instrument with 20 physical items and 9 psychological items.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Healthy Sciences, Granada, Spain